CLINICAL TRIAL: NCT00423085
Title: A 24-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-finding Evaluation of the Efficacy, Safety, and Tolerability of the Once-daily Rivastigmine Transdermal Patch in Patients With Probable Alzheimer's Disease (MMSE 10-20)
Brief Title: Efficacy and Safety of Rivastigmine Transdermal Patch in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CENA713D1301; CENA713D1301E1; NCT00531609 (obsolete NCT alias)
Record Dates: First submitted 2007-01-11; First posted 2007-01-17 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Alzheimer's Disease
Keywords: rivastigmine，Alzheimer's Disease, transdermal patch
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Participants received daily matching placebo patch for the duration of the 24-week double-blind treatment phase of the study.
  Interventions: Drug: Placebo
- rivastigmine 5 cm^2 (Experimental): During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks and thereafter daily rivastigmine 5 cm^2 patch. For patients who experienced intolerability, the dose was adjusted to rivastigmine 2.5 cm^2 daily. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
  Interventions: Drug: Rivastigmine transdermal patch
- Rivastigmine 10 cm^2 (Experimental): During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks, rivastigmine 5 cm^2 patch for the next 4 weeks, rivastigmine 7.5 cm^2 patch for the next 4 weeks and then rivastigmine 10 cm^2 patch for the final 4 weeks. For patients who experienced intolerability, the dose was adjusted downward. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
  Interventions: Drug: Rivastigmine transdermal patch

INTERVENTIONS:
Drug: Rivastigmine transdermal patch — Rivastigmine transdermal patch was provided in the following sizes and doses:
  2.5 cm^2 (4.5 mg), 5 cm^2 (9 mg), 7.5 cm^2 (13.5 mg), and 10 cm^2 (18 mg). The caregiver applied one patch on the back of a patient, placed alternately from the right to the left side at approximately the same time each day.
  Arms: Rivastigmine 10 cm^2; rivastigmine 5 cm^2
Drug: Placebo — Placebo transdermal patch was provided in the following sizes: 2.5 cm^2, 5 cm^2, 7.5 cm^2 and 10 cm^2. The caregiver applied one patch on the back of a patient, placed alternately from the right to the left side at approximately the same time each day.
  Arms: Placebo

SUMMARY:
The purpose of this study was to investigate the 5cm^2 and 10cm^2 doses of rivastigmine transdermal patch in terms of efficacy and safety in patients with probable Alzheimer's Disease (MMSE [Mini Mental State Examination] 10-20). A 52-week extension phase evaluated the safety and tolerability of long-term treatment by rivastigmine transdermal patch in patients with probable Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Patients were randomly assigned in a double-blind manner to one of the 3 treatment arms (placebo, rivastigmine 5 cm^2 and rivastigmine 10 cm^2) in a ratio of 1:1:1. During the Double-blind treatment phase, patients entered a 16-week Titration Period followed by an 8-week Maintenance Period. During the open-label extension phase, all patients started treatment with a 2.5 cm^2 patch and the dose was increased to 10 cm^2 over a 16-week titration period, followed by a maintenance period of 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria
* A clinical diagnosis of probable AD according to NINCDS/ADRDA criteria
* An MMSE score of > or = 10 and < or = 20

Exclusion Criteria:

* A current DSM-IV diagnosis of major depression
* Taken rivastigmine in the past
* A score of > 5 on the Modified Hachinski Ischemic Scale (MHIS) Other protocol-defined inclusion/exclusion criteria may apply

Other protocol-defined inclusion/exclusion criteria may apply

Extension Phase Eligibility Criteria

Inclusion Criteria:

* Patients who have completed the Double-blind Treatment Phase on study medication

Exclusion Criteria

* Patients who have any important protocol deviations until the completion of the Double-blind Treatment Phase

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Hokkaido Region, Hokkaido, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned in a double-blind manner to one of the 3 treatment arms (placebo, rivastigmine 5 cm^2 and rivastigmine 10 cm^2) in a ratio of 1:1:1. Following the 24-week double-blind treatment phase, participants could enroll in the open-label extension phase, where all participants were titrated up to the 10 cm^2 patch dose.
Groups:
- Rivastigmine 5 cm^2: During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks and then daily rivastigmine 5 cm^2 patch. For patients who experienced intolerability, the dose was adjusted to rivastigmine 2.5 cm^2 daily. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
- Rivastigmine 10 cm^2: During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks, rivastigmine 5 cm^2 for the next 4 weeks, rivastigmine 7.5 cm^2 patch for the next 4 weeks and then rivastigmine 10 cm^2 patch for the final 4 weeks. For patients who experienced intolerability, the dose was adjusted downward. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
- Open-label Extension: All participants started treatment with daily rivastigmine 2.5 cm^2 patch. The dose was increased to 5, 7.5, and 10 cm^2 after 4 weeks of treatment at each dose level. One patch was applied once daily. The dose level reached by each individual patient at the end of this 16 weeks was maintained for the rest of the study duration (Maintenance Period). A predetermined "allowed adjustment" scheme was followed in patients who required dose adjustment due to low tolerability.
Period: 24-Week Double-Blind Treatment Phase
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2 | Open-label Extension
Started | 288 | 284 | 287 | 0
Completed | 242 | 220 | 228 | 0
Not Completed | 46 | 64 | 59 | 0
Not completed — Adverse Event | 21 | 38 | 34 | 0
Not completed — Withdrawal by Subject | 8 | 16 | 11 | 0
Not completed — Unsatisfactory therapeutic effect | 7 | 6 | 7 | 0
Not completed — Protocol Violation | 8 | 3 | 7 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: 52-Week Open-Label Extension Phase
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2 | Open-label Extension
Started | 0 | 0 | 0 | 637 (Patients who completed the 24-wk treatment phase were eligible to enroll in the open-label extension)
Completed | 0 | 0 | 0 | 474
Not Completed | 0 | 0 | 0 | 163
Not completed — Adverse Event | 0 | 0 | 0 | 97
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 37
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 18
Not completed — Protocol deviation | 0 | 0 | 0 | 9
Not completed — Death | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2 | Total
Number analyzed (Participants) | 286 | 282 | 287 | 855
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data for the double-blind treatment phase is provided for the safety population. This population consists of all randomized patients who received at least one dose of study medication and had at least one safety assessment after baseline.
  years | 74.5 (7.36) | 74.3 (7.46) | 75.1 (6.85) | 74.6 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 194 | 195 | 584
  Male | 91 | 88 | 92 | 271

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale - Japan Cognitive Subscale (ADAS-J Cog)
Description: The Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) was used to measure change in cognitive function. The ADAS-J cog score ranges from 0-70, with higher total scores indicating more impairment. A negative change score indicates improvement from baseline.
Time Frame: Baseline and Week 24
Population: The Intent-to-treat population: This population includes all randomized patients who received at least one dose of study drug and had at least a baseline and any post-baseline assessment on treatment (i.e. not more than 2 days after the last known date of study drug) for one of the primary efficacy variables. LOCF was utilized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 265 | 266 | 268
units on a scale
  Baseline Score | 24.8 (9.46) | 25.2 (9.62) | 25.0 (9.93)
  Week 24 Score | 26.1 (11.49) | 25.7 (11.70) | 25.1 (11.25)
  Change from Baseline | 1.3 (5.07) | 0.5 (4.96) | 0.1 (5.04)

2. Primary Outcome: Overall Clinical Rating of Change From Baseline to Week 24 Measured by the Clinician's Interview-Based Impression of Change Plus - Japan (CIBIC Plus-J)
Description: The overall clinical rating of change from baseline to week 24 measured by the 7-point CIBIC plus-J scale. The Clinician's Interview-Based Impression of Change plus Caregiver Input consists of 3 subscales: Disability Assessment of Dementia Scale, Behavioral Pathology in Alzheimer's Disease Rating Scale and Mental Function Impairment Scale, as well as the Clinician's Global Impression of Change (CGIC). Participants are scored according to the following:
  1. Markedly improved
  2. Moderately improved
  3. Minimally improved
  4. Unchanged
  5. Minimally worse
  6. Moderately worse
  7. Markedly worse
Time Frame: Baseline and Week 24
Population: Intent-to-treat population utilizing LOCF.
Measure: Number; unit: Participants
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 267 | 269 | 270
Participants
  Markedly improved | 0 | 0 | 0
  Moderately improved | 5 | 12 | 6
  Minimally improved | 36 | 45 | 53
  Unchanged | 111 | 109 | 109
  Minimally worse | 84 | 82 | 78
  Moderately worse | 29 | 21 | 22
  Markedly worse | 2 | 0 | 2

3. Secondary Outcome: Change From Baseline in CIBIC Plus-J Score Disability Assessment for Dementia (DAD)
Description: The Disability Assessment for Dementia (DAD) was used to assess levels of difficulty in activities of daily living (ADL). The DAD is administered through an interview with the caregiver. A total score is obtained by adding the rating for each question and converting this to a total score out of 100 (%). Higher scores represent less disability in ADL while lower scores indicate more dysfunction. A positive change score indicates an improvement from baseline.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. Only patients with a valid baseline and post-baseline score were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 267 | 269 | 269
units on a scale
  Baseline Score | 66.70 (19.902) | 64.19 (20.571) | 64.15 (21.921)
  Week 24 Score | 62.54 (22.395) | 61.19 (22.415) | 62.27 (23.691)
  Change from Baseline | -4.16 (12.443) | -2.99 (10.259) | -1.88 (10.657)

4. Secondary Outcome: Change From Baseline in CIBIC Plus-J Score Behavioral Pathology in Alzheimer's Disease Rating Scale (Behave-AD)
Description: BEHAVE-AD was used to assess patient behavior and psychiatric symptoms. It covers symptoms in seven categories: paranoid and delusional ideation, hallucinations, activity disturbances, diurnal rhythm disturbances, aggressiveness, affective disorders and anxieties, and phobias. Caregivers rate behavioral symptoms on a 0-3 scale. The total score can range from 0 to 66, with a lower score indicating better function. A negative change score indicates an improvement from baseline.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. Only patients with a valid baseline and post-baseline score were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 267 | 269 | 270
units on a scale
  Baseline Score | 4.8 (4.50) | 4.7 (4.96) | 5.4 (5.15)
  Week 24 Score | 4.8 (5.41) | 4.6 (5.03) | 5.1 (5.89)
  Change from Baseline | -0.1 (3.76) | -0.1 (4.17) | -0.3 (4.70)

5. Secondary Outcome: Change From Baseline in CIBIC Plus-J Score Mental Function Impairment Scale (MENFIS)
Description: MENFIS was used to assess patient cognitive and psychiatric function, and evaluates core symptoms of dementia including cognitive, motivational and emotional aspects. The total score ranges from 0 to 78. The higher the score, the greater the functional deficit. A negative change score indicates an improvement from baseline.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. Only patients with a valid baseline and post-baseline score were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 267 | 269 | 270
units on a scale
  Baseline Score | 23.2 (11.13) | 24.3 (11.72) | 24.6 (11.36)
  Week 24 Score | 26.1 (12.68) | 26.5 (13.43) | 26.2 (12.69)
  Change from Baseline | 2.9 (6.18) | 2.2 (5.86) | 1.6 (5.82)

6. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE)
Description: The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. Only patients with a valid baseline and post-baseline score were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rivastigmine 5 cm^2 | Rivastigmine 10 cm^2
Number analyzed (Participants) | 251 | 236 | 246
units on a scale
  Baseline Score | 16.7 (2.87) | 16.9 (2.88) | 16.4 (3.09)
  Week 24 Score | 16.4 (4.21) | 16.6 (4.62) | 16.4 (4.47)
  Change from Baseline | -0.3 (2.82) | -0.3 (3.05) | 0.0 (2.87)

7. Secondary Outcome: Extension Phase: Change From Extension Phase Baseline to End of Extension in Mini-Mental State Examination (MMSE)
Description: The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement. This outcome measured the change in MMSE from the beginning of the open-label extension phase through to Week 52 of the extension phase.
Time Frame: Extension Phase Baseline and Week 52 of extension phase
Population: Intent-to-treat population utilizing last observation carried forward. This population includes all patients who received at least one dose of open-label study medication and had at least one efficacy assessment on treatment in the open-label extension Phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Extension Arm: All participants started treatment with a daily rivastigmine 2.5 cm^2 patch. The dose was increased to 5, 7.5, and then 10 cm^2 after 4 weeks of treatment at each dose level. One patch was applied once daily. The dose level reached by each individual patient at the end of this 16 weeks was maintained for the rest of the study duration (Maintenance Period) for a total of 52 weeks. A predetermined "allowed adjustment" scheme was followed in participants who required dose adjustment due to low tolerability.
Arm/Group | Open-label Extension Arm
Number analyzed (Participants) | 577
units on a scale
  Extension Baseline | 16.6 (4.43)
  End of Extension | 14.9 (5.58)
  Change from Baseline | -1.7 (3.28)

8. Secondary Outcome: Extension Phase: Change From Extension Phase Baseline to End of Extension in CIBIC Plus-J Score Disability Assessment for Dementia (DAD)
Description: The Disability Assessment for Dementia (DAD) was used to assess levels of difficulty in activities of daily living. The DAD is administered through an interview with the caregiver. A total score is obtained by adding the rating for each question and converting this to a total score out of 100 (%). Higher scores represent less disability in activities of daily living while lower scores indicate more dysfunction. A positive change score indicates an improvement from baseline.
Time Frame: Extension Phase Baseline and Week 52 of extension phase
Population: Intent-to-treat population utilizing last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Extension Arm
Number analyzed (Participants) | 567
units on a scale
  Extension Baseline | 61.99 (22.939)
  End of Extension | 51.95 (25.407)
  Change from Baseline | -10.04 (14.089)

9. Secondary Outcome: Extension Phase: Change From Extension Phase Baseline to End of Extension in Modified Crichton Scale
Description: The Modified Crichton Scale includes a total of seven items evaluated in eight grades that assess basic activities of daily living, communication functions, psychiatric symptoms and quality of life; the total score can range from 0 to 56, with a lower score indicating better function. A negative change score indicates an improvement from baseline.
Time Frame: Extension Phase Baseline and Week 52 of extension phase
Population: Intent-to-treat population utilizing last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Extension Arm
Number analyzed (Participants) | 634
units on a scale
  Extension Baseline | 20.0 (10.04)
  End of Extension | 24.0 (11.30)
  Change from Baseline | 4.0 (6.74)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 24-week double-blind treatment phase and during the 52-week open-label extension phase.
Description: Data presented in the Placebo, Rivastigmine 5 cm^2 and Rivastigmine 10 cm^2 columns represent AEs collected during the 24-week double blind treatment phase of the study. Data presented in the Open-Label Extension column are AEs collected during the 52-week open-label extension phase of the study, after completion of the double-blind phase.
Groups:
- Placebo (24 Weeks): Participants received daily matching placebo patch for the duration of the 24-week double-blind treatment phase of the study.
- Rivastigmine 5 cm^2 (24 Weeks): During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks and thereafter daily rivastigmine 5 cm^2 patch. For patients who experienced intolerability, the dose was adjusted to rivastigmine 2.5 cm^2 daily. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
- Rivastigmine 10 cm^2 (24 Weeks): During the 16-week titration period patients received daily rivastigmine 2.5 cm^2 patch for the first 4 weeks, rivastigmine 5 cm^2 patch for the next 4 weeks, rivastigmine 7.5 cm^2 patch for the next 4 weeks and then rivastigmine 10 cm^2 patch for the final 4 weeks. For patients who experienced intolerability, the dose was adjusted downward. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
- Open-Label Extension (52 Weeks): All participants started treatment with daily rivastigmine 2.5 cm^2 patch. The dose was increased to 5, 7.5, and 10 cm^2 after 4 weeks of treatment at each dose level. One patch was applied once daily. The dose level reached by each individual patient at the end of this 16 weeks was maintained for the rest of the study duration (Maintenance Period). A predetermined "allowed adjustment" scheme was followed in patients who required dose adjustment due to low tolerability.
Arm/Group | Placebo (24 Weeks) | Rivastigmine 5 cm^2 (24 Weeks) | Rivastigmine 10 cm^2 (24 Weeks) | Open-Label Extension (52 Weeks)
Serious Adverse Events (participants affected / at risk) | 20/286 | 14/282 | 18/287 | 74/637
Other Adverse Events (participants affected / at risk) | 157/286 | 206/282 | 214/287 | 491/637
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (24 Weeks) (N=286) | Rivastigmine 5 cm^2 (24 Weeks) (N=282) | Rivastigmine 10 cm^2 (24 Weeks) (N=287) | Open-Label Extension (52 Weeks) (N=637)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Condition aggravated (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholangitis suppurative (Infections and infestations) | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 2 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 6
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2 | 2 | 2
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (24 Weeks) (N=286) | Rivastigmine 5 cm^2 (24 Weeks) (N=282) | Rivastigmine 10 cm^2 (24 Weeks) (N=287) | Open-Label Extension (52 Weeks) (N=637)
Constipation (Gastrointestinal disorders) | 12 | 6 | 6 | 43
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 9 | 33
Nausea (Gastrointestinal disorders) | 9 | 3 | 20 | 40
Vomiting (Gastrointestinal disorders) | 11 | 11 | 23 | 58
Application site erythema (General disorders) | 55 | 106 | 113 | 220
Application site oedema (General disorders) | 7 | 35 | 31 | 64
Application site pruritus (General disorders) | 61 | 92 | 100 | 201
Nasopharyngitis (Infections and infestations) | 32 | 22 | 33 | 95
Contusion (Injury, poisoning and procedural complications) | 6 | 9 | 8 | 39
Weight decreased (Investigations) | 4 | 7 | 10 | 35
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 5 | 32
Dermatitis contact (Skin and subcutaneous tissue disorders) | 40 | 69 | 68 | 162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.